CLINICAL TRIAL: NCT04353947
Title: Induction and Recognition of Emotions in Healthy Older Adults, Alzheimer's Disease and Parkinson's Disease
Brief Title: Induction and Recognition of Emotions
Acronym: IRE
Status: Withdrawn | Type: Observational
Why Stopped: COVID 19
Sponsor: University of Valencia (Other)
Collaborators: Asociación Parkinson Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: UV-INV_ETICA-1217558
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Healthy Older Adults; Alzheimer's Disease; Parkinson's Disease
Keywords: Healthy older adults; Alzheimer's disease; Parkinson's disease; Mood induction; Positive emotions; Negative emotions
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy older adults: Healthy older adults with 65 years or older
  Interventions: Diagnostic Test: Mini Cognitive Examination (MCE); Diagnostic Test: Beck Depression Inventory-II (BDI-II); Diagnostic Test: Global Deterioration Scale (GDS); Diagnostic Test: Memory alteration test (M@T); Diagnostic Test: Spanish-Complutense Verbal Learning Test (TAVEC); Diagnostic Test: Barcelona test (BT); Diagnostic Test: Rey-Osterrieth Complex Figure Test (ROCFT); Diagnostic Test: Positive and Negative Affect Scale (PANAS); Diagnostic Test: Auto-Assessment Manikins (SAM)
- Older adults with Alzheimer's disease: Older adults with Alzheimer's disease with 65 years or older
  Interventions: Diagnostic Test: Mini Cognitive Examination (MCE); Diagnostic Test: Beck Depression Inventory-II (BDI-II); Diagnostic Test: Global Deterioration Scale (GDS); Diagnostic Test: Memory alteration test (M@T); Diagnostic Test: Spanish-Complutense Verbal Learning Test (TAVEC); Diagnostic Test: Barcelona test (BT); Diagnostic Test: Rey-Osterrieth Complex Figure Test (ROCFT); Diagnostic Test: Positive and Negative Affect Scale (PANAS); Diagnostic Test: Auto-Assessment Manikins (SAM)
- Older adults with Parkinson's disease: Older adults with Alzheimer's disease with 65 years or older
  Interventions: Diagnostic Test: Mini Cognitive Examination (MCE); Diagnostic Test: Beck Depression Inventory-II (BDI-II); Diagnostic Test: Global Deterioration Scale (GDS); Diagnostic Test: Memory alteration test (M@T); Diagnostic Test: Spanish-Complutense Verbal Learning Test (TAVEC); Diagnostic Test: Barcelona test (BT); Diagnostic Test: Rey-Osterrieth Complex Figure Test (ROCFT); Diagnostic Test: Frontal assessment battery (FAB); Diagnostic Test: Positive and Negative Affect Scale (PANAS); Diagnostic Test: Auto-Assessment Manikins (SAM)

INTERVENTIONS:
Diagnostic Test: Mini Cognitive Examination (MCE) — This test provides information on temporal and spatial orientation, fixation, concentration and calculation, memory and language and construction.
Diagnostic Test: Beck Depression Inventory-II (BDI-II) — This test evaluates the absence or presence of depressive symptoms.
Diagnostic Test: Global Deterioration Scale (GDS) — This scale measures the level of deterioration of the subject.
Diagnostic Test: Memory alteration test (M@T) — In this test different memory subtypes are evaluated.
Diagnostic Test: Spanish-Complutense Verbal Learning Test (TAVEC) — This test is used to assess immediate memory, deferred memory and learning ability.
Diagnostic Test: Barcelona test (BT) — This test evaluates categorical evocation and verbal fluency. The categorical recall subtest consists of recalling the maximum number of words linked to a specific category "animals" in 1 minute. In the case of verbal fluency, the subject is asked to evoke the maximum number of words that begin with the letter "p" in 3 minutes.
Diagnostic Test: Rey-Osterrieth Complex Figure Test (ROCFT) — In this test, the person must carefully copy a complex geometric drawing, which must be memorized later. The first part evaluates multiple cognitive processes such as planning, motor skills, working memory, and visual-constructive and spatial skills. In the second part, memory is evaluated.
Diagnostic Test: Frontal assessment battery (FAB) — This test is a composite tool for assessing executive functions related to the frontal lobe.
  Groups: Older adults with Parkinson's disease
Diagnostic Test: Positive and Negative Affect Scale (PANAS) — It is a self-report questionnaire made up of 20 items (10 of positive affect and another 10 of negative affect) that the subject must answer, obtaining in this way a score in positive affectivity (AP subscale) and another in negative affectivity (AN subscale).
Diagnostic Test: Auto-Assessment Manikins (SAM) — It is a self-report questionnaire that assesses the emotional response of the subject, in this case, through a mood induction task that plays different films scenes.

SUMMARY:
This study evaluates the differences in cognitive function between healthy older adults, older adults with mild Alzheimer's type dementia and older adults with Parkinson's disease and if there are differences in valence assessment and activation that produce them a mood induction task. Subjects are assessed using neuropsychological tests and then a mood induction task based on movie clips is applied.

DETAILED DESCRIPTION:
Different neuropsychological tests will be used to assess the differences in cognitive function in the different groups, whose scores are expected to be lower in the group of older adults with Alzheimer's disease (AD) and older adults with Parkinson's disease (PD).

After studying the cognitive function in the different groups, we proceed to check through a task based on movie clips if there are also differences in the valence assessment (liking/disliking depending on the emotion induced by scenes from different films) and activation (excitement caused by each one of the movie scenes), hoping to find differences for the negative emotions taking into account the cognitive difficulties that both (the EA group and the EP group) may have for processing this type of cognitively more demanding information; instead, it is possible that the positivity effect continues to affect these patients so that for positive emotions there are no differences between the different groups.

ELIGIBILITY:
Inclusion Criteria:

For the group of healthy older adults:

* MEC score greater than 26 points.
* GDS between 1 and 3.

For the mild EA group:

* MEC score between 18 and 23 points.
* GDS between 3 and 4.

For the EP group:

* MEC score greater than 23 points.
* GDS between 1 and 3.
* FAB score equal to or less than 11 points.

General Exclusion Criteria:

Participants cannot have:

* Significant asymptomatic neurovascular disease
* History of previous symptomatic stroke
* Alcohol or drug abuse/dependence
* Severe psychiatric symptoms
* Depressive symptoms higher than mild

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: * Healthy older adults will be recruited from the Third Age Classrooms of the municipality of Quart de Poblet.
  * The older adults with mild Alzheimer's disease will be recruited through the Neurology Department of the General Hospital of Valencia.
  * The older adults with Parkinson's disease will be recruited through the Valencia Parkinson Association.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 5-10 minutes
  This test is evaluated on a maximum of 30 points. Participants with scores equal to or below 23 would be considered cognitively deficient.
Beck Depression Inventory-II (BDI-II) | 5-10 minutes
  In this test, a score of 0-13 indicates absence of depression, 14-19 mild depression, 20-28 moderate depression, and 29-63 severe depression.
Global Deterioration Scale (GDS) | 30 minutes
  This scale indicates seven possible stages: 1. Absence of Cognitive Deficit; 2. Very slight cognitive deficit; 3. Mild Cognitive Deficit; 4. Moderate cognitive deficit; 5. Moderately severe cognitive deficit; 6. Severe cognitive deficit; 7. Very severe cognitive deficit.
Memory alteration test (M@T) | 5-10 minutes
  This cognitive test is evaluated on a maximum of 50 points. The optimal cut-off point for distinguishing mild cognitive impairment of the amnesiac type from subjective memory complaints is 37 points. The optimal cut-off point for Alzheimer's disease is 31 points.
Spanish-Complutense Verbal Learning Test (TAVEC) | 30 minutes
  The evaluator reads a 16-word shopping list in five different essays and in each of them the evaluated person must mention those words that he or she remembers. After 20 minutes, the subject is asked to remember them again.
Barcelona test (BT) | 5 minutes
  In this test, the subject is considered to have a good categorical evocation when he is able to evoke more than 16 animals in 1 minute and a good verbal fluency when he is able to evoke more than 19 words beginning with "p" in 3 minutes.
Rey-Osterrieth Complex Figure Test (ROCFT) | 10 minutes
  The direct score (PD) in the copy of the Rey figure that would leave 50% of the population below is 30 points, while in the reproduction of the Rey figure from memory the PD that would leave 50% below of the population is 21 points.
Frontal assessment battery (FAB) | 10 minutes
  The maximum score to be obtained in this test is 18 points. To consider that the subject presents alterations in the frontal lobe and, therefore, altered executive functions, his score must be equal to or less than 11 points.
Positive and Negative Affect Scale (PANAS) | 10 minutes
  The final score of this scale is the sum of the 10 terms on the positive scale and the sum of the 10 terms on the negative scale, with the value assigned for the responses on the positive scale being positive and negative for the responses on the negative scale.
Auto-Assessment Manikins (SAM) | 5-10 minutes
  This questionnaire measures the valence (liking/disliking depending on the emotion induced by scenes from different movies), the arousal (excitement caused by each of the movie scenes) and mastery or emotional control (self-perception of the control exerted on the environment and the emotion itself).

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Melendez, Psychology, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
All the information of the study, as well as its results, will be shared in scientific publications and conferences related to the research area.
  The information that is intended to be published in scientific journals includes: 1) Study Protocol, 2) Statistical Analysis, 3) Informed Consent Form, 4) Clinical Study Results.

REFERENCES:
- [Result] Fernandez-Aguilar L, Ricarte J, Ros L, Latorre JM. Emotional Differences in Young and Older Adults: Films as Mood Induction Procedure. Front Psychol. 2018 Jul 3;9:1110. doi: 10.3389/fpsyg.2018.01110. eCollection 2018. PMID 30018584
- [Result] Carvalho S, Leite J, Galdo-Alvarez S, Goncalves OF. The Emotional Movie Database (EMDB): a self-report and psychophysiological study. Appl Psychophysiol Biofeedback. 2012 Dec;37(4):279-94. doi: 10.1007/s10484-012-9201-6. PMID 22767079
- [Result] Alves H, Koch A, Unkelbach C. Why Good Is More Alike Than Bad: Processing Implications. Trends Cogn Sci. 2017 Feb;21(2):69-79. doi: 10.1016/j.tics.2016.12.006. Epub 2017 Jan 4. PMID 28063663
- [Result] Alves H, Koch A, Unkelbach C. The differential similarity of positive and negative information - an affect-induced processing outcome? Cogn Emot. 2019 Sep;33(6):1224-1238. doi: 10.1080/02699931.2018.1549022. Epub 2018 Nov 26. PMID 30475089
- [Result] Reed AE, Carstensen LL. The theory behind the age-related positivity effect. Front Psychol. 2012 Sep 27;3:339. doi: 10.3389/fpsyg.2012.00339. eCollection 2012. PMID 23060825
- [Result] Nashiro K, Mather M. Effects of emotional arousal on memory binding in normal aging and Alzheimer's disease. Am J Psychol. 2011 Fall;124(3):301-12. doi: 10.5406/amerjpsyc.124.3.0301. PMID 21977692